CLINICAL TRIAL: NCT06615986
Title: Evaluation of a Human Milk Oligosaccharide-Based Synbiotic Supplement for Intestinal Microbiota Dysbiosis
Brief Title: Human Milk Oligosaccharide-Based Synbiotic Supplement for Intestinal Microbiota Dysbiosis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001729; 001729-H
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Healthy Volunteers
Keywords: Gut Barrier; Intestinal Health; PLASMA LIPIDS; Artherosclerosis; Low-Density Lipoprotein (LDL); Cholesterol; Lipoproteins; Human Milk Oligosaccharides (HMO); Gut Microbiota; Symbiotic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiosyn in Healthy Volunteers (Experimental): Participants will receive 2 doses of Cardiosyn daily by mouth (2 sachets) for a total of 16.2 grams. Each does (sachet) is 8.1 grams.
  Interventions: Dietary Supplement: Cardiosyn

INTERVENTIONS:
Dietary Supplement: Cardiosyn — Two sachets by mouth daily. Each dose (sachet) is 8.1 grams. For 2 doses it will be 16.2 grams per person per day.

SUMMARY:
Background:

Human intestines are home to a complex gut flora, also called microbiome; this is a natural occurring community of bacteria, fungi, yeast, and viruses. Changes in the balances of the gut flora can lead to illnesses, such as diabetes, colorectal cancer, and inflammatory bowel diseases. Synbiotics are dietary supplements people take to maintain proper balances of their gut flora aiming to improve health.

Objective:

To find out if a synbiotic supplement can increase the type and amount of beneficial gut bacteria in healthy people as well as improve cardio-vascular protection markers. The supplement contains a natural sugar from human milk.

Eligibility:

Healthy people aged 18 years or older who eat a typical western diet. They must take no medications (with a few exceptions).

Design:

Participants will have 2 clinic visits.

The first visit will start with screening. They will have a blood test and wait around 2 hours for the results of the blood test. The test will determine if they are eligible for the study.

Eligible participants will have additional blood drawn during the screening visit. They will be given a kit to collect a stool sample at home with instructions. They may complete a 3-day food diary. They will meet with a nutritionist and a physician by phone, telehealth, or in person.

The supplement is a powder that is mixed with water or another noncarbonated drink. Participants will drink 2 doses per day. Each dose will be 1 hour before or after a meal.

The second visit will be about 8 weeks after the first. Participants may repeat the 3-day food diary and nutrition visit. The physical exam, blood tests, and stool sample will be repeated.

DETAILED DESCRIPTION:
Study Description:

This pilot proof-of-principle (PoP) study will investigate mechanisms of action of a human milk oligosaccharide (HMO)-based synbiotic supplement, Cardiosyn (a combination of prebiotics and pro-biotics). Synbiotics for gut microbiota are known to exert multiple beneficial effects, including anti-inflammatory and antioxidant actions, and normalizing blood lipids and iron markers in healthy human subjects.

Objectives:

Primary Objective:

To measure changes in microbiome determined by the increase of the population of Lactobacillus Plantarum and Bifidobacterium Bifidum.

Secondary Objectives:

Measure the level of adherence to the symbiotic supplementation.

Measure the effect of the synbiotic supplementation in plasma.

Measure the effect of synbiotic supplementation on gut integrity.

Tolerability and GI symptoms secondary to gut microbiome changes.

Tertiary/Exploratory Objectives:

Identify possible associations between the gut microbiome change and biomarkers.

Endpoints: Primary Endpoint:

At least an increase in the population of Lactobacillus Plantarum and Bifidobacterium Bifidum.

Secondary Endpoint:

Reported intake by the subject and counting the number of the remaining supplement

Biomarkers such as serum and fecal calprotectin, hs-CRP, serum iron, hepcidin, hemoglobin, lipid profile and TMAO

Measurement of gut integrity marker (serum zonulin) in plasma

Number of participants that tolerated study supplement for full duration of study

Number of participants with GI reported symptoms according to CTCAE v5.0

Tertiary/Exploratory Endpoints:

Measurement of changes of microbiome and biomarkers in plasma (16S RNA microbiota analysis initially with potential for more extensive and novel analysis).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy males and females between the ages 18 to 99.
* Subject understands the protocol and provides written, informed consent in addition to a willingness to comply with specified follow-up evaluations.
* Subjects taking no medications, with a few exceptions (sporadic medication and medications known to not significantly affect the microbiome, per PI discretion).
* Screening labs within normal levels. Deviations of the screening labs from normal levels up to CTCAE v5, grade 1 are allowed per PI discretion.

EXCLUSION CRITERIA:

* Pregnancy or women currently breastfeeding.
* Subjects currently on other prebiotics and/or probiotics supplementation.
* Subjects that are vegetarians or vegans or not on a typical western diet.
* Subjects planning to initiate new medications or already taking medications that may interfere or modify gut microbiome.
* Subjects with allergy or known hypersensitivity to any components of the supplement.
* Subjects with weight changes greater than 20% over the past 3 months.
* Subjects planning a significant change in diet or exercise levels.
* Subjects with chronic diarrhea, gastric bypass or lap-band procedures, ostomies, bowel motility problems, or other known conditions that could affect intestinal fat absorption.
* Anticipated surgery during the study period.
* Any other reason or clinical condition that the Investigators judge would interfere with study participation and/or be unsafe for a participant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Mean change in population of Lactobacillus plantarum and Bifidobacterium bifidum | 8 weeks
  To assess changes in the microbiome, we will measure the increase in the populations of Lactobacillus plantarum and Bifidobacterium bifidum.

SECONDARY OUTCOMES:
Reported intake by the subject and counting the number of remaining supplement | 8 weeks
  Measure adherence to the symbiotic supplementation regimen.
Mean change of biomarkers such as serum and fecal calprotectin, hs-CRP, serum iron, hepcidin, hemoglobin in plasma | 8 weeks
  Assess the effect of synbiotic supplementation on plasma levels.
Fold increase in Lactobacillus or Bifidobacterium over baseline | 8 weeks
  Evaluate the impact of synbiotic supplementation on gut integrity.
Number of participants that tolerated symbiotic supllementation | 8 weeks
  Assess participant tolerabiltiy related to changes in the gut microbiome to synbiotic supplementation for duration of study
Number of gastrointestinal symptoms reported by participants using Common Terminology Criteria for Adverse Events version 5.0 | 8 weeks
  Gastrointestinal symptoms related to changes in the gut microbiome reported by participants using Common Terminology Criteria for Adverse Events version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Amar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting approximately 6 months after publication and available indefinitely.
Access Criteria: Data will be shared through the NHLBI BioData Catalyst, which is a controlled access repository.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001729-H.html